CLINICAL TRIAL: NCT02477449
Title: A Phase I Dose Escalating Study Evaluating the Pharmacokinetics, Tolerability and Safety of Istaroxime Infusion for 24 Hours in Chinese Healthy Volunteers
Brief Title: Istaroxime Infusion for 24 Hours in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: CVie Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVie2015001
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: safety; istaroxime
MeSH Terms: interventions — Istaroxime; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- low dose group (Experimental): 8 subjects in 0.25ug/kg/min group were administrated Istaroxime + 0.9% NS; All the subjects were given infusion of study drugs for 24 hours, and then were observed for 48 hours in the clinic.
  Interventions: Drug: istaroxime
- mid dose group (Experimental): 12 subjects in 0.5ug/kg/min group randomly received Istaroxime placebo + 0.9% NS (2 subjects), 0.9% NS alone (2 subjects) and Istaroxime + 0.9% NS (8 subjects). All the subjects were given infusion of study drugs for 24 hours, and then were observed for 48 hours in the clinic.
  Interventions: Drug: istaroxime; Drug: 9% Saline (NS)
- high dose group (Experimental): 12 subjects in 1.0 ug/kg/min group randomly received Istaroxime placebo + 0.9% NS (2 subjects), 0.9% NS alone (2 subjects) and Istaroxime + 0.9% NS (8 subjects). All the subjects were given infusion of study drugs for 24 hours, and then were observed for 48 hours in the clinic.
  Interventions: Drug: istaroxime; Drug: 9% Saline (NS)

INTERVENTIONS:
Drug: istaroxime — 8 subjects in 0.25ug/kg/min group were administrated Istaroxime + 0.9% NS fo12 subjects in 0.5ug/kg/min or 1.0 ug/kg/min group randomly received Istaroxime placebo + 0.9% NS (2 subjects), 0.9% NS alone (2 subjects) and Istaroxime + 0.9% NS (8 subjects).
Drug: 9% Saline (NS) — infusion for 24 hours
  Arms: high dose group; mid dose group

SUMMARY:
Phase 1 study to investigate safety of istaroxime in healthy chinese volunteers.

DETAILED DESCRIPTION:
32 subjects (F: M=1:1) were randomized in three dose groups (0.25-0.5-1.0ug/kg/min). 8 subjects in 0.25ug/kg/min group were administrated Istaroxime + 0.9% NS; 12 subjects in 0.5ug/kg/min or 1.0 ug/kg/min group randomly received Istaroxime placebo + 0.9% NS (2 subjects), 0.9% NS alone (2 subjects) and Istaroxime + 0.9% NS (8 subjects). All the subjects were given infusion of study drugs for 24 hours, and then were observed for 48 hours in the clinic. At least 1 week should be kept between two dose groups. Escalation to the higher dose will occur after the lower dose group has been completed and no significant safety issues are found.

ELIGIBILITY:
Inclusion Criteria:

1. Age at 18-45 years (inclusive)
2. Male or Non-pregnant, non-lactating women
3. Chinese healthy subjects
4. Body mass index (BMI) at 19-24 kg/m2 (inclusive) and body weight at 50-100kg
5. Lab examinations (include but not limited: Hemoglobin, white blood cell counting, differential count, creatinine,Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT),Total bilirubin and urinalysis) are within normal range or out of normal range but no clinical significance.
6. Vital signs in screening phase: SBP100-139mmHg, DBP 50-89 mmHg, pulse rate 45-90 bpm. Holter is within normal range or out of normal range but no clinical significance.
7. Both physical examination and ECG at baseline are normal or abnormal but no clinical significance
8. Women of childbearing age during the trial must be willing to use a medically acceptable method of contraception, which include surgical sterilization (tubal ligation / hysterectomy), and double barrier methods of hormonal contraception.
9. Subjects well communicate with investigators, understanding the requirements of investigators and being willing to sign the ICF before conducting any study-related procedure.
10. Subjects are willing to stay at the phase I ward throughout the study.

Exclusion Criteria:

1. Disease history in liver, kidney, endocrine, cardiovascular, neurological, psychiatric, gastrointestinal tract, lungs, immune, skin, blood, or metabolic disorders or cancer, that may have great impact on the study results.
2. Presence of pancreatitis, intestinal obstruction, glaucoma, prostatic hypertrophy, adrenal disease, hyperthyroidism or gallbladder disease (subjects had experienced cholecystectomy will not be excluded)
3. History of clinical significant disease in the past 4 weeks before screening visit
4. Presence of diseases which are known to disturb the absorption, distribution, metabolism or excretion of Istaroxime
5. Physical examinations, medical history, ECG, vital signs or lab examination are deemed to be abnormal and clinical significant
6. Be intolerant or allergy to Istaroxime, lactose or any similar substances
7. Significantly abnormal diets are conducted within 4 weeks before screening visit
8. Blood donation or loss equal to or exceeds 400ml in the past 6 months
9. Participating in the any other drug study in the past 3 months
10. Administrated OTC drugs including vitamin supplements and herbal (Occasional use of paracetamol will not be excluded)
11. Regular use of any prescription drug (Hormonal birth control pills or hormone replacement therapy will not be excluded)
12. Drinking beverage or eat food containing caffeinated / xanthine or poppy seed since 48 hours before study drugs administration; or drinking beverage or eat food containing grapefruit, oranges or Chinese tea 14 days before the study drug administration
13. Receiving the therapy of drugs including cytochrome P450 3A4 or cytochrome P450 2C8 inhibitors or inducers (eg barbiturates, carbamazepine, erythromycin, phenytoin, thiazoline TZDs, Rifampin)
14. Women at Lactation period or with positive pregnancy test
15. Tongue piercing or lip piercing occurred 30 days before the study drug administration
16. Smoke or tobacco is used 60 days before the study drug administration
17. History of abusing any substance including infusion drugs, alcohol and opium
18. Positive alcohol breathing test within 1day or drink alcohol within 1week
19. Abusing drugs (include Opioids, oxycodone, methamphetamine, amphetamine, cannabinoids, cocaine, barbiturates, benzodiazepines class, methadone, buprenorphine and phencyclidine)
20. History of heart disease
21. Planning to be pregnant in the recent 3 months
22. Participating any other interventional strudy in the past 30 days
23. History of bronchial asthma or blood porphyria disease
24. HbsAg, anti-HCV, anti-HIV or anti - syphilis are positive
25. Holter examination is abnormal and clinical significant
26. Subjects are not eligible for the study judged by investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
safety of istaroxime in healthy volunteers is measured by varition of heart functon, blood pressure and heart ratio | one week
  safety of istaroxime in healthy volunteers is measured by

CONTACTS AND LOCATIONS:
Locations (1):
- The 307th hospital of chinese People's liberation army, Beijing, China